CLINICAL TRIAL: NCT07371195
Title: Relationship Between Upper Cervical Mobility and Temporomandibular Joint Range of Motion in Patients With Temporomandibular Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Other Study IDs: Upper Cervical Mobility
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Temporomandibular Disorders (TMD); Temporomandibular Joint Dysfunction Syndrome; Cervicogenic Headache
Keywords: Temporomandibular Joint; Temporomandibular Disorders; Upper Cervical Spine; Cervical Mobility
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome; Post-Traumatic Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Temporomandibular Disorder Group: Fifty patients with temporomandibular disorder will undergo evaluation of upper cervical spine mobility (flexion, extension, and rotation) and TMJ range of motion (opening, lateral excursion, and protrusion) using standardized instruments (CROM device and ruler/caliper).

SUMMARY:
Upper cervical spine mobility plays a crucial role in temporomandibular joint (TMJ) function. This observational study investigates the relationship between upper cervical spine mobility and TMJ range of motion in patients diagnosed with temporomandibular disorders (TMD). Cervical hypomobility may restrict mandibular movement and contribute to TMJ dysfunction through shared biomechanical and neuromuscular mechanisms.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are multifactorial conditions involving the temporomandibular joint, masticatory muscles, or both. Prior research indicates a strong association between TMD and cervical spine dysfunction, with patients frequently exhibiting neck pain, reduced cervical motion, and muscular tenderness.

This study explores how upper cervical mobility (flexion, extension, and rotation) correlates with TMJ range of motion (mouth opening, lateral excursion, and protrusion). The aim is to identify whether cervical spine hypomobility contributes to restricted jaw movement in TMD patients.

A total of 50 participants with TMD will undergo standardized clinical measurements of cervical mobility using a CROM device and TMJ motion using a ruler or caliper. Pearson or Spearman correlation coefficients will be applied to evaluate the association between cervical and TMJ movement parameters.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable individuals who consent to participate in the study.
* Age between 18 and 50 years.
* Both male and female participants.
* Patients diagnosed with temporomandibular joint (TMJ) dysfunction for at least three months.

Exclusion Criteria:

* Presence of systemic diseases.
* Body mass index (BMI) greater than 30 kg/m².
* Pregnancy.
* Recent physical therapy for cervical spine disorders, headaches, or temporomandibular dysfunction.
* Cervical radiculopathy or other neurological disorders.
* History of trauma or major psychological problems.
* Generalized joint hypermobility.
* Down syndrome.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be adult patients (both male and female) aged 18 to 50 years who have been clinically diagnosed with temporomandibular joint (TMJ) dysfunction for more than three months. All participants will be recruited from the outpatient clinic of the Faculty of Physical Therapy, Deraya University, Minya, Egypt. Eligible participants will be medically stable and free from systemic or neurological disorders that could affect cervical or temporomandibular mobility.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Upper Cervical Spine Mobility | Single assessment session (baseline only)
  Upper cervical spine mobility (flexion, extension, and left and right rotation) will be measured in degrees using a CROM device. Participants will be seated in an upright position, and each movement will be measured twice following standardized procedures. The mean value of both readings will be used for analysis.
Temporomandibular Joint Range of Motion (TMJ ROM) | Single assessment session (baseline only)
  TMJ range of motion will be measured in millimetres using a standard ruler or digital calliper. Measurements include maximum mouth opening, lateral excursion (left and right), and protrusion. Each measurement will be taken twice, and the average will be recorded in millimetres to ensure reliability.
Correlation Between Upper Cervical Mobility and TMJ Range of Motion | Single assessment session (baseline only)
  The relationship between upper cervical spine mobility (measured in degrees using the CROM device) and TMJ range of motion (measured in millimetres using a ruler or calliper) will be analysed statistically. Pearson or Spearman correlation coefficients will be applied, depending on data normality, to determine the strength and direction of association.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Deraya University, Minya, Menia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No